CLINICAL TRIAL: NCT03490474
Title: Pain Modulatory Profiles in Massage for Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB201800213
Record Dates: First submitted 2018-03-21; First posted 2018-04-06 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Healthy; Musculoskeletal Pain
Keywords: conditioned pain modulation (CPM); diffuse noxious inhibitory control (DNIC); massage; hypoalgesia
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pain Inducing Massage (Experimental): Participants will receive manual pressure applied to one myofascial trigger point.
  Interventions: Other: Pain Inducing Massage
- Pain Free Massage (Active Comparator): Participants will receive light touch applied to one myofascial trigger point.
  Interventions: Other: Pain Free Massage
- Coldpressor (Placebo Comparator): Participants will place hand into water cooled to 6 degrees Celsius (males) or 8 degrees Celsius (females).
  Interventions: Other: Coldpressor

INTERVENTIONS:
Other: Pain Inducing Massage — Participants will receive 60 seconds of manual pressure applied to one myofascial trigger point so the participant rates the pain = 5/10 on a scale from 0 to 10. This will be followed by 30 seconds of complete pressure release. This will occur 4 times.
  Arms: Pain Inducing Massage
Other: Pain Free Massage — Participants will receive 60 seconds of light touch applied to one myofascial trigger point so the participant rates the pain = 0/10 on a scale from 0 to 10. This will be followed by 30 seconds of complete pressure release. This will occur 4 times.
  Arms: Pain Free Massage
Other: Coldpressor — Participants will place their non-dominant hand into water cooled by a refrigeration unit temperature of 6 degrees Celsius (males) or 8 degrees Celsius (females). The participant will place his or her hand in the cooled water for 60 seconds followed by a 30 second break in which the participant will remove his or her hand from the water. This will occur 4 times.
  Arms: Coldpressor

SUMMARY:
One in ten adults experience widespread pain. Neck pain, for example, is a prevalent condition with a high rate of recurrence that affects between 10.4% and 21.3% of the population annually.

Massage is a common manual therapy intervention for individuals with musculoskeletal pain. However, the mechanisms of massage are not well established. Also, the conditioned pain modulation (CPM) paradigm is a dynamic quantitative sensory testing measure of a pain inhibitory process in which pain sensitivity is lessened in response to a remotely applied painful stimulus.

This study will evaluate the association between pain inducing massage and the conditioned pain modulation paradigm.

DETAILED DESCRIPTION:
Conditioned pain modulation (CPM) is the physical manifestation of the diffuse noxious inhibitory control (DNIC), an endogenous pain inhibitory pathway in which pain inhibits pain. Conditioned pain modulation is less efficient in individuals with chronic pain conditions and it is a predictor for the development of chronic pain.

Massage is a common manual therapy intervention for individuals with musculoskeletal pain. Greater changes in pain sensitivity occur following pain inducing massage suggesting a mechanism dependent upon the efficiency of the conditioned pain modulation response.

The study team will evaluate the association between pain inducing massage and the conditioned pain modulation paradigm. Healthy participants will be randomly assigned to receive a pain inducing massage, a pain free massage, or participate in a coldpressor task. Pre-and post intervention pain sensitivity including conditioned pain modulation will be assessed. The study team will determine if analgesia induced by massage is similar to the conditioned pain modulation paradigm and compare changes in pain sensitivity between groups.

Previous research has indicated pain inducing massage is more effective than pain free massage suggesting a mechanism dependent upon conditioned pain modulation. However, this study will be the first to systematically investigate if analgesia induced by pain inducing massage is similar to the conditioned pain modulation paradigm. Furthermore, this study will be the first to determine the association between baseline conditioned pain modulation and massage related hypoalgesia.

ELIGIBILITY:
Inclusion Criteria:

* pain free
* blood pressure under 140/90 mmHg
* ability of therapist to locate necessary trigger points on participant

Exclusion Criteria:

* blood pressure over 140/90 mmHg
* inability of therapist to locate necessary trigger points on participant
* systemic medical condition known to affect sensation (i.e. diabetes)
* regular use of prescription pain medication to manage pain
* current or history of chronic pain condition
* currently using blood thinning medication
* any blood clotting disorder such as hemophilia
* any contraindication to application of ice or cold pack, such as: uncontrolled hypertension, cold urticaria, cryoglobulinemia, paroxysmal cold hemoglobinuria, and circulatory compromise
* non-English speaking

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Pressure Pain Threshold | 2 hours
  Pressure in kilograms at which ascending pressure stimulus first changes from pressure to painful

SECONDARY OUTCOMES:
Change from baseline in Thermal Pain Threshold and Tolerance | 2 hours
  Temperature at which ascending thermal stimulus first changes from warm to painful and maximum temperature tolerated
Change from baseline in Pressure Pain Tolerance | 2 hours
  Pressure in kilograms at which ascending pressure is no longer tolerated
Change from baseline in Ramp and Hold | 2 hours
  Participants will rate their pain using a 101 point mechanical visual analog scale to thermal stimuli of 45, 47, 49, and 50 degree Celsius each of 5 seconds duration will be applied to the forearm and to the muscle on the side of the neck
Change from baseline in Temporal Summation | 2 hours
  Participants will rate their pain using a 0 to 10 numeric rating scale to a train of 10 50 degree Celsius heat pulses will be applied to the skin in the plantar surface of the hand.
Change from baseline in Conditioned Pain Modulation | 2 hours
  Pressure in kilograms at which ascending pressure stimulus applied to the foot first changes from pressure to painful both prior to and immediately following immersion of the opposite hand in a cold water bath

CONTACTS AND LOCATIONS:
Overall Officials: Joel Bialosky, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No